CLINICAL TRIAL: NCT00327808
Title: Multi-Center, Randomized, Double-Blind, Repeated Doses Study to Evaluate the Safety, Tolerability and Pharmacodynamic Activity of Inhaled TPI-1020 Versus Inhaled Budesonide in Smokers With Mild Reversible Asthma
Brief Title: Inhaled TPI-1020 Versus Inhaled Budesonide in Smokers With Mild Reversible Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPI 1020-202
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: Smokers; Adults; Inflammatory markers
MeSH Terms: conditions — Asthma | interventions — NCX 1020; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaler (Experimental): TPI 1020
  Interventions: Drug: TPI-1020
- Inhaler cortico. (Active Comparator): Budesonide inhaler
  Interventions: Drug: budesonide

INTERVENTIONS:
Drug: TPI-1020 — 600 mcg BID x 14 days followed by 1200 mcg BID x 7 days
  Arms: Inhaler
Drug: budesonide — 400 mcg BID x 14 days then 800 mcg/day x 7 more days
  Arms: Inhaler cortico.

SUMMARY:
The investigators will look at TPI-1020 safety and tolerability in mild to moderate asthmatic smoker subjects.

DETAILED DESCRIPTION:
This study will assess and compare the safety and tolerability of inhaled TPI 1020 versus budesonide. Pharmacokinetic (PK) and pharmacodynamic (PD) parameters will also be studied in a sub-group of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 through 65 years of age.
* Smoking history of more than 5 pack/years but less than 25 pack/years and who have no desire to quit smoking despite physician's advice and who currently smoke at least 5 cigarettes per day.
* Mild to moderate, stable, allergic asthma as defined by American Thoracic Society (ATS) criteria 1
* History of episodic wheeze and shortness of breath
* Subjects currently and only receiving inhaled short-acting bronchodilator treatment for asthma.

Exclusion Criteria:

* History or symptoms of significant autoimmune, hematological, or neurological disease, including transient ischemic attack (TIA), stroke, seizure disorder, or behavioural disturbances that are judged clinically significant by the Investigator
* History of serious adverse reaction or hypersensitivity to corticosteroids
* Abnormal chest X-ray that is judged clinically significant
* Pregnant or lactating or have positive plasma pregnancy test
* Use of oral/parenteral/inhaled corticosteroids within the last 28 days or injectable depot corticosteroids within the last 6 weeks.
* Use of any other asthma-related medications within 1 month of Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of multiple doses of TPI-1020 in subjects with asthma who smoke | 22 days

SECONDARY OUTCOMES:
To compare sputum neutrophil and eosinophil counts on Day 0 versus Day 15 and Day 22 | 22 days
To determine pharmacodynamic effects on forced expiratory volume in 1 second (FEV1) over 8 hours on Day 1 and Day 14 | 22 days
To compare pre-dose FEV1 measurements on multiple days throughout the study | 22 days
To compare peak flow measurements throughout the study | 22 days
To compare the use of daily rescue medication (salbutamol) throughout the study | 22 days
To determine the plasma pharmacokinetic (PK) profile on a sub-group of subjects on the first and last day of the dosing period | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Renzi, MD, Study Director — Syntara
Locations (7):
- Canada (7):
  - McMaster University Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - CARL, Laval, Quebec
  - Montreal Chest Institute, Montreal, Quebec
  - Hopital Sacre Coeur, Montreal, Quebec
  - Centre Hospitalier St-Sacrement, Ste-Foy, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de l'Hopital Laval, Ste-Foy, Quebec